CLINICAL TRIAL: NCT04992182
Title: Reactogenicidad, Seguridad e Inmunogenicidad de Dosis de Refuerzo de Vacunas Contra SARS-CoV-2 en Chile (Estudio REFUERZO)
Brief Title: Reactogenicity, Safety, and Immunogenicity of Covid-19 Vaccine Booster
Acronym: REFUERZO
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Universidad del Desarrollo (Other)
Collaborators: Ministry of Health, Chile (Other Government); University of Chile (Other); Pontificia Universidad Catolica de Chile (Other)
Responsible Party: Principal Investigator, Rafael Araos, Assistant Professor of Medicine, Principal Investigator, Universidad del Desarrollo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2021-71
Record Dates: First submitted 2021-08-02; First posted 2021-08-05 (Actual); Last update posted 2021-08-05 (Actual); Status verified 2021-08

CONDITIONS: Covid19
Keywords: covid-19; inactivated vaccine; booster; Chile
MeSH Terms: conditions — COVID-19 | interventions — sinovac COVID-19 vaccine; BNT162 Vaccine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Inactivated vaccine booster (Experimental): One standard IM CoronaVac dose (0.5 mL)
  Interventions: Biological: Inactivated vaccine booster
- mRNA vaccine booster (Experimental): One standard IM BNT162b2 dose (0.3 mL)
  Interventions: Biological: mRNA vaccine booster
- Viral vector vaccine booster (Experimental): One standard IM ChAdOx1 dose (0.5 mL)
  Interventions: Drug: Viral vector vaccine booster
- Placebo (Placebo Comparator): Saline solution IM (0.3 mL)
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Placebo — 0.3 mL IM saline solution
  Arms: Placebo
Biological: Inactivated vaccine booster — 0.5 mL IM
  Other Names: CoronaVac
  Arms: Inactivated vaccine booster
Biological: mRNA vaccine booster — 0.3 mL IM
  Other Names: BNT162b2
  Arms: mRNA vaccine booster
Drug: Viral vector vaccine booster — 0.5 mL IM
  Other Names: ChAdOx1
  Arms: Viral vector vaccine booster

SUMMARY:
Preliminary data suggest that inactivated vaccine-induced neutralizing antibodies against SARS-CoV-2 decrease at six months after vaccination. Observational, unpublished data also indicate that vaccine effectiveness against Covid-19 wanes over time. Thus, the investigators aimed to determine the reactogenicity, safety, and immunogenicity of a homologous or heterologous booster of SARS-CoV-2 vaccines among people already immunized with an inactivated SARS-CoV-2 vaccine. The study focuses on the elderly population and healthcare workers.

ELIGIBILITY:
Inclusion Criteria:

* Full immunization with CoronaVac (2 doses; 0,28) prior to April 15, 2021
* Being a resident of any of the eligible Nursing Homes (located in the Metropolitan Region of Chile)
* Healthcare workers of one of the eligible Nursing Homes.
* Healthcare workers of Hospital de Urgencia Asistencia Publica (HUAP, Santiago, Chile)

Exclusion Criteria:

* Prior history of Covid-19
* Not able to consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 534 (Actual)
Dates: Start 2021-07-08 (Actual); Primary Completion 2021-08-31 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
Early humoral response | Baseline (90-120 days after second dose of CoronaVac) and 15 days post booster dose
  Change in SARS-CoV-2 neutralizing antibody levels
Immunogenicity | Baseline, 15, 30, 60, and 90 days post booster dose
  Change in SARS-CoV-2 neutralizing antibody levels

SECONDARY OUTCOMES:
Reactogenicity | days 7, 28, and 3 months post booster dose
  Solicited and unsolicited. Events will be assessed by scheduled visits performed by nursing home´s nurse stuff. Telephone numbers, including the PI´s cell phone will be available 24/7 for reporting any unsolicited reaction. Reporting will follow national regulations available at the Institute of Public Health web page (https://www.ispch.cl/anamed/farmacovigilancia/vacunas/como-notificar-esavi/)
Safety of booster dose | In addition to the scheduled visits mentioned in Outcome 3, Telephone numbers, including the PI´s cell phone will be available 24/7 throughout the study (1 year) for reporting any unsolicited reaction.
  Number of subjects presenting serious adverse events post booster dose.

CONTACTS AND LOCATIONS:
Locations (2):
- Chile (2):
  - ELEAMs (Nursing Homes), Santiago
  - Hospital de Urgencia Asistencia Publica, Santiago

IPD SHARING:
Plan to Share IPD: No
Owing to data privacy regulations, the individual-level data in this study cannot be shared (Law N19.628).